CLINICAL TRIAL: NCT00969904
Title: Double Blind, Randomized, Placebo-controlled, Two-way Crossover, Pilot Study to Assess the Effect of High Dose N-acetylcysteine on Small Airways and on Inflammation and Oxidative Stress in COPD Patients.
Brief Title: Pilot Study to Assess the Effect of High Dose N-acetylcysteine (NAC) in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Wilfried De Backer, MD PhD, University Hospital, Antwerp
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PML_DOC_0804; EC 8/40/128
Record Dates: First submitted 2009-08-31; First posted 2009-09-01 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2012-06

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: N-acetylcysteine
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: N-acetylcysteine — 600 mg TID for 12 weeks
  Arms: 1
Drug: placebo — placebo tablet TID for 12 weeks
  Arms: 2

SUMMARY:
Studies suggest that N-acetylcysteine (NAC) potentially reduces inflammation and hyperinflation in patients with COPD.

In this pilot study the efficacy, safety and tolerability of high dose NAC in 12 patients with moderate COPD will be examined. These patients will receive a placebo for 12 weeks and NAC for 12 weeks in a dosage of 3 times 600 mg a day on top of their usual medication in a randomized crossover design. All subjects will be followed for 28 weeks.

The effect of high dose NAC on small airways will be assessed by measuring the total and peripheral airway resistance calculated with Computational Fluid Dynamics (CFD). The effect on oxidative stress will be assessed by measuring exhaled NO and specific markers (CRP, erythrocyte sedimentation rate, IL-6, 8-isoprostane, H2O2, TNF-alfa, glutathione, GPX, SOD and IL-8) in blood and Exhaled Breath Condensate (EBC). Dynamic and static lung volumes will be assessed by spirometry, body plethysmography and diffusion. Quality of life and symptoms will be assessed by the St George Respiratory Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with documented COPD based on the following criteria:

   * Smoking history of at least 10 pack-years
   * Decreased Tiffeneau index (FEV1/(FVC < 0.70)
2. Patients aged ≥ 40 years
3. Patients who stopped smoking since more than 1 month
4. Patients who present moderate COPD with an FEV1 between 50 and 80% of predicted (GOLD 2)
5. Patients should be treated according to GOLD guidelines

Exclusion Criteria:

1. Unstable patients who developed an exacerbation during the last 8 weeks
2. Patients who are current smokers or stopped less than 1 month
3. Patients who are allergic to acetylcysteine or to another element of the product
4. Patients with phenylketonuria or an untreated active peptic ulcer
5. Patients with any stage kidney and/or heart insufficiency or hypertension
6. Patients already treated with NAC for more than 6 months or during the last 3 months
7. Patients on continuous treatment with oral, inhalation, intravenous or intramuscular corticosteroids
8. Patients who are pregnant or are breast-feeding
9. Patients who are treated with orally administered cephalosporins
10. Patients using supplements containing antioxidants as vitamins C or E

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-03; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To assess the effect of high dose NAC (1800 mg)on small airways by measuring the total and peripheral airway resistance calculated with CFD | at baseline, after 12 weeks of placebo and after 12 weeks of NAC
To assess the effect of high dose NAC (1800 mg)on oxidative stress by measuring exhaled NO and oxidative stress markers in blood and EBC | at baseline, after 12 weeks of placebo and after 12 weeks of NAC.

SECONDARY OUTCOMES:
To assess dynamic and static lung volumes by spirometry, body plethysmography and diffusion | will be assessed at all visits
To assess quality of life by the SGRQ | will be assessed at all visits
To assess the tolerability and safety of high dose NAC | all visits

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried A De Backer, MD, PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- University Hospital Antwerp, Edegem, Antwerp, Belgium

REFERENCES:
- [Derived] De Backer J, Vos W, Van Holsbeke C, Vinchurkar S, Claes R, Parizel PM, De Backer W. Effect of high-dose N-acetylcysteine on airway geometry, inflammation, and oxidative stress in COPD patients. Int J Chron Obstruct Pulmon Dis. 2013;8:569-79. doi: 10.2147/COPD.S49307. Epub 2013 Nov 22. PMID 24293993